CLINICAL TRIAL: NCT00160810
Title: Outcome Study of Complex Distal Radius Fractures: Open Reduction Internal Fixation (ORIF) With A Volar Fixed Angled Plate Versus A Distal Radius Volar (DRV) Plate Versus External Fixation
Brief Title: Outcome Study of Complex Distal Radius Fractures
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 86-2001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2012-06

CONDITIONS: Distal Radius Fractures
Keywords: distal; radius; fractures
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect information about how people do after different treatments of a broken wrist to see if one treatment has better results.

DETAILED DESCRIPTION:
Complex distal radius fractures are a common problem treated by orthopaedic surgeons. The purpose of this study is to compare the outcome between complex distal radius fractures treated with open reduction and internal fixation using a volar fixed angled plate versus and external fixator versus DRV. The hypothesis is that the volar fixed angled plate will have a superior outcome both radiographically and clinically.

ELIGIBILITY:
Inclusion Criteria:

* distal radius fracture

Exclusion Criteria:

* none

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic clinic
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2001-04; Primary Completion 2010-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Wrist Range of Motion | one year post-op
  An improvement of all aspects of wrist motion (extension, flexion, supination and pronation) over one year post-op.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) and Patient Rated Wrist Evaluation (PRWE) scores | one year post-op
  An improvement of the DASH and PRWE scores over one year post-op.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Wright, M.D., Principal Investigator — University of Florida
Locations (1):
- UF and Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States